CLINICAL TRIAL: NCT06533696
Title: A Comparison of Microscopy and Enzyme Linked Immunosorbent Assay for Diagnosis of Giardia Lamblia in Children, Sohag
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Arwa youssif Abdelsabor, demonstrator at medical parasitology department at faculty of medicine sohag, Sohag University
Other Study IDs: Soh-Med-24-06-21MS
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Giardia Lamblia Infection
MeSH Terms: conditions — Giardiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- immunocompromised: immunocompromised cancer, renal failure and undernourished patients
- immunocompetent: exclude cancer, renal failure patients

SUMMARY:
The present study was done to evaluate the efficacy of Human anti Giardia lamblia antibody (ELISA) kitst in comparison to direct microscopy in the diagnosis of G. lamblia in stool specimens from immunocompetent and immunocompromised children with diarrhea and other gastrointestinal symptoms.

DETAILED DESCRIPTION:
Giardia duode- nalis is an intestinal protozoan parasite with a worldwide distribu- tion in human and

animals ( Dixon BR.,2021)

According to WHO reports in 2010, giardiasis is estimated to cause approximately 28.2 million cases of

diarrhea (WHO.,2015)

The prevalence of giardiasis is 2 to 5% in developed countries and 20 to 30% in developing countries in children (Luis et al.,2017)

The fecal-oral route is the main transmission mode of G. duodenalis . Drinking water, food and

vegetables contaminated by G. duodenalis cysts are the main sources of transmission ( Adam Rodney.,2021)

The common clinical manifestations of giardiasis include greasy diarrhea (steatorrhea), nausea,

vomiting, abdominal bloating, cramps, malabsorption and weight loss (Taghipour et al .,2022)

The detection and diagnosis of giardiasis present challenges for physicians, especially in regions distant

from high-prevalence areas where a substantial number of asymptomatic patients further complicate

prevalence determination. Symptoms, which closely mimic those of other parasitic diseases, can

confound clinicians, potentially leading to the prescription of ineffective remedies (Escobedo .et al .,2018)

Several different diagnostic systems have been described for the diagnosis of giardiasis: among them are

microscopic diagnosis, molecular methods, and immunoassays such as ELISA for the detection

of Giardia antigen or anti-Giardia antibodies, and Direct Fluorescence Antibody (DFA) test, which

detects antigens present on the cell wall of Giardia cysts ( Sadaka et al .,2015)

The early accurate diagnosis of giardiasis is important for the successful treatment and prevention of

diseases. The routine laboratory diagnosis is performed for the detection of trophozoites or cysts by

microscopic examination of at least three stool samples collected independently (.Uehlinger et al.,2017)

This diagnosis depends upon the times of sampling, patient compliance, application of concentration

methods, and the expertise of the technologists. Furthermore, in recent years, other methods, such as

ELIZA and molecular techniques are used mainly for diagnostic or research purposes. The sensitivity

and specificity of all diagnostic methods can be improved by including alternative diagnostic procedures

that are more rapid and reliable ( Kosack et al.,2017)

The recently licensed commercially available enzyme-linked immunosorbent assay (ELISA) kits are

found to be rapid and effective methods to diagnose Giardia infection in patients with gastrointestinal

symptomatology by detecting G. lamblia associated antigens in stool (Jahan et al.,2014)

ELIGIBILITY:
Inclusion Criteria:

* Immunocompetent and immunocompromised children with diarrhea and other gastrointestinal symptoms with any age and sex group

Exclusion Criteria:

* patients taking anti parasitic treatment within the previous two weeks of stool sample collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Immunocompetent and immunocompromised children with diarrhea and other gastrointestinal symptoms with any age and sex group
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
A Comparison of Microscopy and Enzyme Linked Immunosorbent Assay for Diagnosis of Giardia lamblia in Children, Sohag | 1 year
  evaluate the efficacy of Human anti Giardia lamblia antibody (ELISA) kitst in comparison to direct microscopy in the diagnosis of G. lamblia in stool specimens from immunocompetent and immunocompromised children with diarrhea and other gastrointestinal symptoms.